CLINICAL TRIAL: NCT01392625
Title: A Phase I/II, Randomized Pilot Study of the Comparative Safety and Efficacy of Transendocardial Injection of Autologous Mesenchymal Stem Cells Versus Allogeneic Mesenchymal Stem Cells in Patients With Non-ischemic Dilated Cardiomyopathy.
Brief Title: PercutaneOus StEm Cell Injection Delivery Effects On Neomyogenesis in Dilated CardioMyopathy (The POSEIDON-DCM Study)
Acronym: PoseidonDCM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Sponsor- Investigator; Director of ISCI, Chief Science Officer, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20100968; 1R01HL110737-01 (NIH)
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Non-ischemic Dilated Cardiomyopathy
Keywords: Non ischemic dilated cardiomyopathy; Dilated cardiomyopathy; Heart failure; Cardiac Stem Cell Transplantation; Stem Cells
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Autologous hMSCs (Active Comparator): Group 1 (18 patients) Eighteen (18) patients will be treated with Auto-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Interventions: Biological: Autologous hMSCs
- Allogeneic hMSCs (Active Comparator): Group 2 (18 patients) Eighteen (18) patients will be treated with allogeneic hMSCs (Allo-hMSCs): 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Interventions: Biological: Allogeneic hMSCs

INTERVENTIONS:
Biological: Autologous hMSCs — Cells will be administered via the Biosense Webster MyoStar NOGA Injection Catheter System will be tested in 18 patients via transendocardial injection:
  Group 1 (18 patients) Eighteen (18) patients will be treated with Auto-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Other Names: Biosense Webster MyoStar NOGA Injection Catheter System.
  Arms: Autologous hMSCs
Biological: Allogeneic hMSCs — Cells will be administered via the Biosense Webster MyoStar NOGA Injection Catheter System will be tested in 18 patients via transendocardial injection:
  Group 2 (18 patients) Eighteen (18) patients will be treated with Allo-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Other Names: Biosense Webster MyoStar NOGA Injection Catheter System.
  Arms: Allogeneic hMSCs

SUMMARY:
The technique of transplanting progenitor cells into a region of damaged myocardium, termed cellular cardiomyoplasty1, is a potentially new therapeutic modality designed to replace or repair necrotic, scarred, or dysfunctional myocardium2-4. Ideally, graft cells should be readily available, easy to culture to ensure adequate quantities for transplantation, and able to survive in host myocardium; often a hostile environment of limited blood supply and immunorejection. Whether effective cellular regenerative strategies require that administered cells differentiate into adult cardiomyocytes and couple electromechanically with the surrounding myocardium is increasingly controversial and recent evidence suggests that this may not be required for effective cardiac repair. Most importantly, transplantation of graft cells should improve cardiac function and prevent adverse ventricular remodeling. To date, a number of candidate cells have been transplanted in experimental models, including fetal and neonatal cardiomyocytes5, embryonic stem cell-derived myocytes6, 7, tissue engineered contractile grafts8, skeletal myoblasts9, several cell types derived from adult bone marrow10-15, and cardiac precursors residing within the heart itself16. There has been substantial clinical development in the use of whole bone marrow and skeletal myoblast preparations in studies enrolling both post-infarction patients, and patients with chronic ischemic left ventricular dysfunction and heart failure. The effects of bone-marrow derived mesenchymal stem cells (MSCs) have also been studied clinically.

Currently, bone marrow or bone marrow-derived cells represent highly promising modality for cardiac repair. The totality of evidence from trials investigating autologous whole bone marrow infusions into patients following myocardial infarction supports the safety of this approach. In terms of efficacy, increases in ejection fraction are reported in the majority of the trials.

Non-ischemic dilated cardiomyopathy is a common and problematic condition; definitive therapy in the form of heart transplantation is available to only a tiny minority of eligible patients. Cellular cardiomyoplasty for chronic heart failure has been studied less than for acute MI, but represents a potentially important alternative for this disease.

DETAILED DESCRIPTION:
This is a Pilot Study, intended as a safety assessment prior to a full comparator study. In this Pilot Study, cells administered via the Biosense Webster MyoStar NOGA injection catheter system will be tested in 36 patients in two groups:

Group 1 (18 patients) Eighteen (18) patients will be treated with Auto-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 X 108 (100 million) Auto-hMSCs.

Group 2 (18 patients) Eighteen (18) patients will be treated with Allo-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 X 108 (100 million) Auto-hMSCs.

The first three (3) patients in each group (Group 1 and Group 2) will not be treated less than 5 days apart and will each undergo full evaluation for 5 days to demonstrate there is no evidence of a procedure induced myocardial infarction or myocardial perforation prior to proceeding with the treatment of further patients.

Patients will be randomized in a 1:1 ratio to one of the two groups.

Treatment Strategies: Autologous hMSCs vs. Allogeneic hMSCs. The Study Team will record and maintain a detailed record of injection locations.

If a patient is randomized to Groups 1 (Auto-hMSCs) and the Auto-hMSCs do not expand to the required dose of 1 X 108 cells, each injection will contain the maximum number of cells available.

The injections will be administered transendocardially during cardiac catheterization using the Biosense Webster MyoStar NOGA Catheter System.

For patients randomized to Group 1(Auto-hMSCs); the cells will be derived from a sample of the patient's bone marrow (obtained by iliac crest aspiration) approximately 4-6 weeks prior to cardiac catheterization. For patients randomized to Group 2 (Allo- hMSCs), the cells will be supplied from an allogeneic human mesenchymal stem cell source manufactured by the University of Miami. The Allo-hMSCs for patients in group 2 will be administered after all baseline assessments are completed with an expected range of 2 - 4 weeks post-randomization.

Following cardiac catheterization and cell injections, patients will be hospitalized for a minimum of 2 days then followed at 2 weeks post-catheterization, and at month 2, 3, 6, and 12 to complete all safety and efficacy assessments.

ELIGIBILITY:
Major Inclusion Criteria:

* Be ≥ 18 and < 95 years of age.
* Provide written informed consent.
* Diagnosis of nonischemic dilated cardiomyopathy.
* Be a candidate for cardiac catheterization within 5 to 10 weeks of screening.
* Been treated with appropriate maximal medical therapy for heart failure.
* Ejection fraction below 40% and either a left ventricular end diastolic diameter (LVEDD) > 5.9cm in male subjects, an LVEDD of > 5.6cm in female subjects or left ventricular end diastolic volume index > 125 mL/m2
* Be able to undergo an MRI or CT.

Major Exclusion Criteria:

* Baseline glomerular filtration rate equal or < 45 ml/min/1.73m2.
* Be eligible for or require standard-of-care surgical or percutaneous intervention for the treatment of nonischemic dilated cardiomyopathy.
* Presence of a prosthetic aortic valve or heart constrictive device.
* Presence of a prosthetic mitral valve.
* Previous myocardial infarction (MI) as documented by a clinical history that will include an elevation of cardiac enzymes and/or ECG changes consistent with MI.
* Diagnosis of nonischemic dilated cardiomyopathy due to valvular dysfunction, mitral regurgitation, tachycardia, or myocarditis.
* Previous treatment for post-infarction left ventricular dysfunction including PCI and thrombolytic therapy.
* Documented presence of a known LV thrombus, aortic dissection, or aortic aneurysm.
* Documented presence of epicardial stenosis of 70% or greater in one or more major epicardial coronary arteries.
* Documented presence of aortic stenosis (aortic stenosis graded as 1.5cm2 or less).
* Documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥+2).
* Evidence of a life-threatening arrhythmia in the absence of a defibrillator (nonsustained ventricular tachycardia ≥ 20 consecutive beats or complete second or third degree heart block in the absence of a functioning pacemaker) or QTc interval > 550 ms on screening ECG.
* AICD firing in the past 30 days prior to the procedure
* Be eligible for or require coronary artery revascularization.
* Diabetic with poorly controlled blood glucose levels and/or evidence of proliferative retinopathy.
* Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
* Have liver dysfunction, as evidenced by enzymes (ALT and AST) greater than three times the ULN.
* Have a coagulopathy condition = (INR > 1.3) not due to a reversible cause.
* Known, serious radiographic contrast allergy.
* Known allergies to penicillin or streptomycin.
* Organ transplant recipient.
* Have a history of organ or cell transplant rejection
* Clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Non-cardiac condition that limits lifespan to < 1 year.
* On chronic therapy with immunosuppressant medication.
* Serum positive for HIV, hepatitis BsAg, or viremic hepatitis C.
* Female patient who is pregnant, nursing, or of child-bearing potential and not using effective birth control.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams AR, Trachtenberg B, Velazquez DL, McNiece I, Altman P, Rouy D, Mendizabal AM, Pattany PM, Lopera GA, Fishman J, Zambrano JP, Heldman AW, Hare JM. Intramyocardial stem cell injection in patients with ischemic cardiomyopathy: functional recovery and reverse remodeling. Circ Res. 2011 Apr 1;108(7):792-6. doi: 10.1161/CIRCRESAHA.111.242610. Epub 2011 Mar 17. PMID 21415390
- [Background] Trachtenberg B, Velazquez DL, Williams AR, McNiece I, Fishman J, Nguyen K, Rouy D, Altman P, Schwarz R, Mendizabal A, Oskouei B, Byrnes J, Soto V, Tracy M, Zambrano JP, Heldman AW, Hare JM. Rationale and design of the Transendocardial Injection of Autologous Human Cells (bone marrow or mesenchymal) in Chronic Ischemic Left Ventricular Dysfunction and Heart Failure Secondary to Myocardial Infarction (TAC-HFT) trial: A randomized, double-blind, placebo-controlled study of safety and efficacy. Am Heart J. 2011 Mar;161(3):487-93. doi: 10.1016/j.ahj.2010.11.024. PMID 21392602
- [Background] Hare JM, DiFede DL, Rieger AC, Florea V, Landin AM, El-Khorazaty J, Khan A, Mushtaq M, Lowery MH, Byrnes JJ, Hendel RC, Cohen MG, Alfonso CE, Valasaki K, Pujol MV, Golpanian S, Ghersin E, Fishman JE, Pattany P, Gomes SA, Delgado C, Miki R, Abuzeid F, Vidro-Casiano M, Premer C, Medina A, Porras V, Hatzistergos KE, Anderson E, Mendizabal A, Mitrani R, Heldman AW. Randomized Comparison of Allogeneic Versus Autologous Mesenchymal Stem Cells for Nonischemic Dilated Cardiomyopathy: POSEIDON-DCM Trial. J Am Coll Cardiol. 2017 Feb 7;69(5):526-537. doi: 10.1016/j.jacc.2016.11.009. Epub 2016 Nov 14. PMID 27856208
- [Derived] Premer C, Wanschel A, Porras V, Balkan W, Legendre-Hyldig T, Saltzman RG, Dong C, Schulman IH, Hare JM. Mesenchymal Stem Cell Secretion of SDF-1alpha Modulates Endothelial Function in Dilated Cardiomyopathy. Front Physiol. 2019 Sep 24;10:1182. doi: 10.3389/fphys.2019.01182. eCollection 2019. PMID 31616309
- [Derived] Tompkins BA, Rieger AC, Florea V, Banerjee MN, Natsumeda M, Nigh ED, Landin AM, Rodriguez GM, Hatzistergos KE, Schulman IH, Hare JM. Comparison of Mesenchymal Stem Cell Efficacy in Ischemic Versus Nonischemic Dilated Cardiomyopathy. J Am Heart Assoc. 2018 Jul 12;7(14):e008460. doi: 10.1161/JAHA.117.008460. PMID 30005555
- [Derived] Mushtaq M, DiFede DL, Golpanian S, Khan A, Gomes SA, Mendizabal A, Heldman AW, Hare JM. Rationale and design of the Percutaneous Stem Cell Injection Delivery Effects on Neomyogenesis in Dilated Cardiomyopathy (the POSEIDON-DCM study): a phase I/II, randomized pilot study of the comparative safety and efficacy of transendocardial injection of autologous mesenchymal stem cell vs. allogeneic mesenchymal stem cells in patients with non-ischemic dilated cardiomyopathy. J Cardiovasc Transl Res. 2014 Dec;7(9):769-80. doi: 10.1007/s12265-014-9594-0. Epub 2014 Oct 30. PMID 25354998
- See also: Interdisciplinary Stem Cell Institute University of Miami — http://isci.med.miami.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous hMSCs: Group 1 (18 patients) Eighteen (18) patients will be treated with Auto-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Autologous hMSCs: Cells will be administered via the Biosense Webster MyoStar NOGA Injection Catheter System will be tested in 18 patients via transendocardial injection:
  Group 1 (18 patients) Eighteen (18) patients will be treated with Auto-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
- Allogeneic hMSCs: Group 2 (18 patients) Eighteen (18) patients will be treated with allogeneic hMSCs (Allo-hMSCs): 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
  Allogeneic hMSCs: Cells will be administered via the Biosense Webster MyoStar NOGA Injection Catheter System will be tested in 18 patients via transendocardial injection:
  Group 2 (18 patients) Eighteen (18) patients will be treated with Allo-hMSCs: 20 million cells/ml delivered in a dose of 0.5 ml per injection x 10 injections for a total of 1 x 108 (100 million) Auto-hMSCs.
Period: Overall Study
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Started | 18 | 19
Completed | 16 | 18
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous hMSCs | Allogeneic hMSCs | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.0) | 54.4 (11.5) | 55.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 11 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 10 | 15 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Participants Injection status in the trial [Count of Participants; unit: Participants]
  No | 2 | 1 | 3
  Yes | 16 | 18 | 34
Participants Ejection Fraction % in the trial [Mean (Standard Deviation); unit: percentage] | 21.7 (6.2) | 22.5 (6.5) | 22.1 (6.3)
Enrollment End Diastolic diameter (CM) [Mean (Standard Deviation); unit: centimeters] | 7.0 (1.6) | 7.2 (1.2) | 7.1 (1.4)
New York Heart Association Class [Count of Participants; unit: Participants] — Population: 37 participants were randomized to treatment numbers and assignments but 3 did not continue with treatment and not included in the analysis.
  Participants
    number analyzed (Participants) | 16 | 18 | 34
    Class I - no limitation | 6 | 4 | 10
    Class II - Slight Limitation of Physical Activity | 8 | 9 | 17
    Class III - Marked Limitation of Physical Activity | 2 | 5 | 7
    Class IV -Inability to carry on physical activity | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Treatment-emergent Serious Adverse Events (TE-SAEs)
Description: Incidence of TE-SAEs is defined as the composite of: death, non-fatal MI, stroke, hospitalization for worsening heart failure, cardiac perforation, pericardial tamponade, sustained ventricular arrhythmias (characterized by ventricular arrhythmias lasting longer than 15 seconds or with hemodynamic compromise), or any other potential late effects detected and corroborated by clinical presentation, laboratory investigations, image analysis and when necessary with biopsy from suspected target sites in the body.
Time Frame: One month post-catheterization
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 16 | 18
Participants
  Upper respiratory tract infection | 1 | 0
  Ventricular tachycardia | 0 | 1
  Device Pacing issue | 0 | 1

2. Secondary Outcome: Measurement of Changes in Peak VO2
Description: Measurement of Peak oxygen consumption (Peak VO2) by treadmill determination during the 12 month follow-up period.
Time Frame: Baseline, 6 month and 12 month
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 16 | 18
ml/kg/min
  Peak VO2 (Baseline) | 16.0 (5.13) | 17.9 (5.17)
  Peak VO2 (6 months) | 15.5 (6.62) | 17.6 (3.55)
  Peak VO2 (1 year) | 16.4 (3.92) | 20.1 (5.10)

3. Secondary Outcome: Measurement of Changes in 6 Minute Walk
Description: Measurement of Six-minute walk test during the 12 month follow-up period
Time Frame: Baseline, 6 month and 12 month
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 16 | 18
meters
  6 minute walk (Baseline) | 416.4 (105.74) | 427.2 (67.35)
  6 minute walk (6 months) | 384.2 (106.96) | 438.7 (106.53)
  6 minute walk (1 year) | 32.3 (12.71) | 35.1 (13.59)

4. Secondary Outcome: Measurement of Changes in Global Ejection Fraction
Description: Measurement of regional left ventricular function, end diastolic and end systolic volume, measured by MRI, and or CT, and echocardiogram.
Time Frame: Baseline, 6 month and 12 month
Measure: Mean (Standard Deviation); unit: % ratio of the SV to Global EDV
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 16 | 18
% ratio of the SV to Global EDV
  Global ejection fraction (Baseline) | 25.2 (10.49) | 37.6 (9.03)
  Global ejection fraction (1 year) | 32.3 (12.71) | 35.1 (13.59)

5. Secondary Outcome: Measurement of Changes in New York Heart Association (NYHA)
Description: Measurement of New York Heart Association (NYHA) functional class during the 12 month follow-up period.
Time Frame: Baseline, 6 month and 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 18 | 19
Participants
  NYHA Class 1 (Baseline) | 6 | 4
  NYHA Class 2 (Baseline) | 8 | 9
  NYHA Class 3 (Baseline) | 2 | 5
  NYHA Class 1 (6 month) | 8 | 12
  NYHA Class 2 (6 month) | 6 | 4
  NYHA Class 3 (6 month) | 1 | 1
  NYHA Class 1 (12 month) | 7 | 14
  NYHA Class 2 (12 month) | 2 | 1
  NYHA Class 3 (12 month) | 2 | 0

6. Secondary Outcome: Measurement of Changes in Minnesota Living With Heart Failure (MLHF) Questionnaire
Description: Measurement of Minnesota Living with Heart Failure (MLHF) Questionnaire during the 12 month follow-up period. It measures the effects of symptoms, functional limitations, and psychological distress on an individual's quality of life. The response scale for all 21 items on the MLHF is based on a 6-point. The Maximum possible scores being 126 and the minimum 0. Higher scores indicate a worse or worsening quality of life, while lower scores or decreasing scores indicate a better quality of life.
Time Frame: Baseline, 6 month and 12 month
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
Number analyzed (Participants) | 16 | 18
scores on a scale
  MLHF (Baseline) | 30.5 [5.0 to 80.0] | 38.0 [10.0 to 82.0]
  MLHF (6 month) | 35 [0.0 to 87.0] | 18 [0.0 to 68.0]
  MLHF (12 month) | 9.0 [0.0 to 41.0] | 12.0 [0.0 to 51.0]

ADVERSE EVENTS:
Time Frame: These AE's were collected over a period of 1 year from the subject signing the consent form.
Arm/Group | Autologous hMSCs | Allogeneic hMSCs
All-Cause Mortality (participants affected / at risk) | 2/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 6/18 | 6/19
Other Adverse Events (participants affected / at risk) | 4/18 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous hMSCs (N=18) | Allogeneic hMSCs (N=19)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — 1-month SAE
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) — 1-month sae
Device Pacing issue (Product Issues) | 0 (0) | 1 (1) — 1-month SAE
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) — 6-month SAE
Cardiac failure (Cardiac disorders) | 2 (3) | 1 (1) — 6-month SAE
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) — 6-month SAE
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — 6-month SAE
Gatrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) — 6-month SAE
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) — 6-month SAE
Subdural heamatoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — 6-month SAE
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — 6-month SAE
Device pacing issues (Product Issues) | 0 (0) | 1 (1) — 6-month SAE
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 6-month SAE
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — 6-month SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous hMSCs (N=18) | Allogeneic hMSCs (N=19)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Treatment Emergent Adverse event at one-month
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) — Treatment Emergent AE at 1-month
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Chest Discomfort (General disorders) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) — Treatment emergent adverse event at 1 month
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Weight increased (Investigations) | 2 (2) | 0 (0) — Treatment emergent adverse event at 1 month
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Migraine (Nervous system disorders) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Device pacing issue (Product Issues) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Treatment emergent adverse event at 1 month
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Treatment emergent adverse event at 1 month
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1) — Treatment emergent adverse event at 1 month

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes